CLINICAL TRIAL: NCT03737162
Title: Bare-metal Stent vs Covered Stent in Chinese Patients With Subclavian Occlusive Lesions: Prospective, Multiple Center, Randomized, Open, Positive Controlled Trail
Brief Title: Bare-metal Stent vs Covered Stent in Chinese Patients With Subclavian Occlusive Lesions
Acronym: BASELINE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Peking University First Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); Shanghai Zhongshan Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Changzheng Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Yong-Quan Gu, Prof., Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: china subclavian
Record Dates: First submitted 2018-11-06; First posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Subclavian Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Covered stent group (Experimental): Covered stent
  Interventions: Procedure: Stent implantation of subclavian artery
- Bare-metal stent group (Active Comparator): Bare-metal stent
  Interventions: Procedure: Stent implantation of subclavian artery

INTERVENTIONS:
Procedure: Stent implantation of subclavian artery — Stent implantation of subclavian artery

SUMMARY:
Bare-metal stent vs Covered stent with subclavian occlusive lesions to verify the efficacy and safety.Study Design are prospective, multiple center, randomized, open, positive controlled, non-inferiority trail.Case total numbers enrollment predict 408 cases，each group 204 cases.Follow up period for 1 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥50 years，sex unlimited；
2. Left subclavian artery disease；
3. The cause of clinical considerations is arteriosclerosis ；
4. The presence of target organ ischemic symptoms, ie dizziness, headache, transient ischemic attack (TIA), stroke, or other related neurological symptoms caused by ischemia of the vertebral artery in the past 6 months, or the presence of arterial stenosis beyond the upper extremity limb ischemia symptoms subclavian；
5. The patient understands the trial objective, understands and accepts the duration of the study，is able and willing to comply with all requirements，including follow-up and evaluation of it, voluntarily participates in the study and signs Informed Consent Form.

   Anatomy Criteria
6. Subclavian artery independent disease（Do not merge carotid or vertebral artery disease ）；
7. Subclavian artery satisfies one of the following criteria：

   1. a) Ultrasonography suggests stenosis ≥ 70%，or CT ANGIOGRAM / angiography showed stenosis ≥ 70%；
   2. Iconography examination confirmed vertebral artery steals；
   3. Length of lesion is not involved in vertebral artery opening；
   4. Lesions in subclavian artery the beginning portion；
8. The stent can reach the site of lesion smoothly as expected.

Exclusion Criteria:

1. Patients with anesthesia contraindications；
2. Serious ipsilateral stroke occurred in the past and may confuse the judgment of the study endpoint ；
3. Patients with severe dementia ；
4. Patients with spontaneous intracerebral hemorrhage in the past 12 months ；
5. Patients stroke episodes recently， CT or MRI suggested that the lesion is large，and may be with the risk of hemorrhagic transformation ；
6. Large size of cerebral infarction or myocardial infarction occurred within 30 days ；
7. Patients with large intracranial aneurysms (diameter> 5mm)，and cannot be treated in advance or contemporaneous ；
8. Chronic total occlusion without obvious cerebral ischemia symptoms ；
9. Patients with hemorrhagic transformation of cerebral arterial thrombosis within 60 days before surgery ；
10. Hemoglobin <100 g/l， Platelet count <125×109/L， INR>1.5， Bleeding time > 1 min，patients with exceeding the upper limits of normal，or heparin-related thrombocytopenia ；
11. Patients unable to perform normal angiographic evaluation or unsafe percutaneous puncture poin；
12. Patients with neurologic disorder that caused transient or permanent neurological deficits within 2 years before the surgery and can not be identified with TIA or stroke ；
13. Patients with other cardiac emboli sources, such as left ventricular aneurysm, intraluminal filling defect, cardiomyopathy, aortic or mitral prosthetic heart valve, calcific aortic stenosis, infective endocarditis, mitral stenosis, atrial septal defect, atrial septal aneurysm, or left atrial myxoma；
14. Surgical contraindications or patients with high risk of surgery defined as having any of the following；It is known that two or more proximal or main coronary artery stenosis ≥70%, untreated or unable to pass；Ejection fraction <30% or New York Heart Association (NYHA) functional class III or higher；Unstable angina，ie angina at resting state and electrocardiogram changes；Currently waiting main organ transplants (ie heart, lung, liver, kidney), or are doing relevant evaluate；Malignant tumor or respiratory insufficiency, life expectancy < 5 years or FORCED EXPIRATORY VOLUME AT ONE SECOND < 30% (predicted)；Dialysis-dependent renal failure； Need to perform other general anesthesia during the same period ；
15. There may be one or more anatomical conditions affecting the normal operative approach in patients； there may be one or more anatomic situations to increase the risk of adverse events in patients with high operative risk；including： Neck radiation therapy history； Radical neck surgery history；Subclavian artery dissection；Lesions series；Severe long segment calcification of the subclavian artery and severe stenosis or occlusion of the basilar artery；Inaccessible lesions by endoluminal methods (Severe distortion of the aortic arch branch, no suitable introduction of arteries, aortic arch anatomy special）；
16. Investigators consider the patient inappropriate to participate in this clinical trial；
17. Those who participated in clinical trials of other drugs or medical devices before the inclusion did not reach the end of the time limit.
18. Rheumatic immune diseases, such as Takayasu arteritis.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2018-04-02 (Actual); Primary Completion 2020-04-03 (Estimated); Study Completion 2020-07-03 (Estimated)

PRIMARY OUTCOMES:
target lesion patency rate（%） | 1 years
  12-month target lesion patency rate（%）

SECONDARY OUTCOMES:
Surgery success rate | 1 day
  Surgery success rate
Rate of complications | 30 days
  Rate of complications within 30 days；
Incidence of myocardial infarction | 30 days
  Incidence of myocardial infarction at 30 days follow up；
Ipsilateral stroke and death rates | 30 days
  Ipsilateral stroke and death rates at 30 days follow up；
Bilateral stroke and death rates | 30 days
  Bilateral stroke and death rates at 30 days follow up；
Subclavian artery restenosis rate | 6、12 months
  Subclavian artery restenosis rate at 6、12 months follow up；
Incidence of composite endpoints of myocardial infarction, stroke, and any death | 30days
  Incidence of composite endpoints of myocardial infarction, stroke, and any death at 30 days
Incidence of composite endpoints of myocardial infarction, stroke, and any death | 6 months
  Incidence of composite endpoints of myocardial infarction, stroke, and any death at 6 months
Incidence of composite endpoints of myocardial infarction, stroke, and any death | 12 months
  Incidence of composite endpoints of myocardial infarction, stroke, and any death at 12 months
Surgical time | Through hospital stay，an average of 10 days
  Surgical time
Hospitalization days | Through hospital stay，an average of 10 days
  Hospitalization days
Hospitalization fees | Through hospital stay，an average of 10 days
  Hospitalization fees

CONTACTS AND LOCATIONS:
Overall Officials: YongQuan Gu YQ Gu, Prof., Principal Investigator — Xuanwu Hospital, Beijing
Locations (6):
- China (6):
  - Peking hospital first University, Beijing
  - The first affiliated Hospital of Dalian Medical University, Dalian
  - Shanghai Changhai Hospital, Shanghai
  - Shanghai Changzheng Hospital, Shanghai
  - Zhongshan Hospital affiliated to Fudan University, Shanghai
  - The first affiliated Hospital of Xi ' an Jiaotong University, Xi'an

IPD SHARING:
Plan to Share IPD: Undecided